CLINICAL TRIAL: NCT02129010
Title: The Pathogenesis of Terson Syndrome and the Role of CSF Tau / Amyloid-ß 40 and 42 in Patients With Aneurysmatic Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Holger Joswig (Other)
Collaborators: Innogenetics N.V., Belgium (Unknown)
Responsible Party: Sponsor-Investigator, Holger Joswig, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: ICPTS-Sma-2012
Record Dates: First submitted 2014-04-27; First posted 2014-05-01 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Subarachnoid Hemorrhage; Terson Syndrome; CSF-proteines
Keywords: subarachnoid hemorrhage; terson syndrome; CSF-proteines; phospho-tau; beta-amyloid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subarachnoid hemorrhage with and without Terson syndrome: Patients with aneurysmatic subarachnoid hemorrhage with and without Terson syndrome

SUMMARY:
Prospective clinical study to investigate the pathogenesis of Terson syndrome and the prognostic value of the CSF-biomarkers tau-protein and amyloid-β 40 and 42 in patients with aneurysmatic subarachnoid hemorrhage. Our two hypotheses are as follows:

1. The incidence of Terson syndrome correlates with the initial intracranial opening pressure (measured with extra ventricular drain)
2. The CSF-biomarkers correlate with the outcome assessed at discharge, 3-, 6- and 12-months postictally using Glasgow-Outcome-Scale-Extended (GOSE) and Euro-Qol-5 as well as with complications related to aneurysmatic subarachnoid hemorrhage such as cerebral vasospasm, delayed cerebral ischemia and re-bleed.

DETAILED DESCRIPTION:
In this prospective clinical study the pathogenesis of Terson syndrome and the prognostic value of the CSF-biomarkers tau-proteine and amyloid-β 40 and 42 in patients with aneurysmatic subarachnoidal hemorrhage are investigated. Intracranial opening pressure will be measured in patients requiring CSF-diversion for acute hydrocephalus and correlated with the incidence of Terson syndrome tested by an opthalmologic exam (group A: Terson syndrome positive, group B: Terson syndrome negative). CSF samples from external ventricular drainages are obtained at day 0, 2 and 6 and concentration of tau-protein and amyloid-β 40 and 42 are determined and correlated to secondary outcome measures such as delayed cerebral ischemia, clinical vasospasm, re-bleed, necessity for surgical intervention secondary to raised intracranial pressure or CSF-diversion. Outcome in terms of Glasgow-Outcome-Scale-Extended and Euro-Qol-5 will be assessed at 3, 6 and 12 months.

CSF from patients undergoing diagnostic or therapeutic tapping of their internal ventricles for normal pressure hydrocephalus or shunt diagnostics serve as a reference for CSF-biomarkers concentration in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* diagnosis of subarachnoid hemorrhage secondary to an intracranial aneurysm
* aneurysmatic subarachnoid hemorrhage must be the principal diagnosis for hospitalization
* an intracranial aneurysm must be confirmed by imaging (Computed tomography, magnet resonance tomography or angiography)
* Patients requiring diagnostic/therapeutic tapping of their internal ventricles for CSF-diversion (shunt) for normal pressure hydrocephalus or shunt diagnostics serve as a control group
* informed consent

Exclusion Criteria:

* younger than 18 years
* other diagnosis such as traumatic or perimesencephalic subarachnoid hemorrhage without an intracranial aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with aneurysmatic subarachnoid hemorrhage requiring CSF-diversion and/or intracranial pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure (ICP) in mmH20 | after insertion of EVD or ICP-probe (between day 0 and 3)
  Initial ICP is measured in mmH20 after insertion of EVD with a riser tube or after insertion of an ICP-probe.

SECONDARY OUTCOMES:
Concentration of CSF-protein phospho-tau | Day 0, 2, 6
  Concentration of CSF-protein phospho-tau taken from EVD-CSF
Concentration of CSF-protein amyloid-ß 40/42 | Day 0, 2, 6
  Concentration of CSF-protein phospho-tau taken from EVD-CSF
Delayed cerebral ischemia | Daily for the duration of hospital stay, an expected average of 3 to 5 weeks
  For the duration of their hospital stay (which can be expected to be an average of 3 to 5 weeks for SAH patients), occurrence of delayed cerebral schema, diagnosed by CT or MRI, is noted (number of patients of cohort).
Clinically manifest vasospasm | Daily for the duration of hospital stay, an expected average of 3 to 5 weeks
  For the duration of their hospital stay (which can be expected to be an average of 3 to 5 weeks for SAH patients), occurrence of clinically manifest vasospasm is noted (number of patients of cohort). Screening will be performed daily by transcranial doppler and confirmation of diagnosis done by CTA or angiography.
Re-bleed | Daily for the duration of hospital stay, an expected average of 3 to 5 weeks
  For the duration of their hospital stay (which can be expected to be an average of 3 to 5 weeks for SAH patients), occurrence of an intracranial re-bleed, diagnosed by CT or MRI, is noted (number of patients of cohort).
Surgery for refractory ICP (decompressive hemicraniectomy) | Daily for the duration of hospital stay, an expected average of 3 to 5 weeks
  For the duration of their hospital stay (which can be expected to be an average of 3 to 5 weeks for SAH patients), the need for surgery for refractory ICP (decompressive hemicraniectomy) is noted (number of patients of cohort). Indication for surgery is made by the treating staff consultant based on ICP, CPP and clinical status.
Necessity of CSF-shunt | Daily for the duration of hospital stay, an expected average of 3 to 5 weeks
  For the duration of their hospital stay (which can be expected to be an average of 3 to 5 weeks for SAH patients), the need for permanent CSF-diversion is noted (number of patients of cohort). Indication for permanent CSF-diversion (usually a ventriculoperitoneal shunt) is made by the treating staff consultant based on radiographic and clinical signs of hydrocephalus secondary to SAH.
Opthalmologic exam | Day 0 to 3; before discharge if initial exam negative
  Occurrence of Terson syndrome is assessed by fundoscopy with chemically dilated pupils (number of patients of cohort).
  Intraocular pressure (mmHg) is measured.

OTHER OUTCOMES:
Glasgow-Outcome-Scale-Extended (GOSE) | initial, 3, 6, 12 months after SAH
  Health outcome is assessed by the study physicians or a study nurse using the Glasgow-Outcome-Scale-Extended (GOSE) with the help of family members if necessary.
Life quality (Euro-Qol-5) | initial, 3, 6, 12 months after SAH
  Life quality is assessed by the study physicians or a study nurse using the Euro-Qol-5 questionnaire with the help of family members if necessary.
Neuropsychological deficits | On day 14 and at 3 and 12 months
  The Montreal Cognitive Assessment (MoCA) is performed at day 14 days. A neuropsychological assessment by a neuropsychologist will then be performed at 3 and 12 months after SAH and includes a combination of the following tests: Alertness (Testbatterie zur Aufmerksamkeitsprüfung, TAP 2.2), Go/Nogo (TAP 2.2), Geteilte Aufmerksamkeit (TAP 2.2), Deux Barrage (2002), Farbe-Wort-Interferenztest (FWIT, after J.R. Stroop, 1985), Regensburger Wortflüssigkeitstest (RWT (2000)), 5-Punkte-Test (HAMASCH, H5PT-R), Frontal Assessment Battery Bedside (FAB), Verbaler Lern- und Merkfähigkeitstest (VLMT), Rey Complex Figure Test (RCFT (1995)), Tiere-Wörter-Test of the test battery Consortium to Establish A Registry for Alzheimer (CERAD), Boston Naming Test (CERAD), Mini-Mental-Status-Examination (CERAD), Trail-Making-Test A (CERAD) and B (CERAD), S-Wörter-Test (CERAD), Apraxie-Prüfung (Goldenberg). Patients' cognitive status is graded as no (regular), or as minimal, moderate or severely disabled.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Joswig, M.D., Principal Investigator — Cantonal Hospital St. Gallen, Dept. of Neurosurgery
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

REFERENCES:
- [Derived] Joswig H, Fournier JY, Hildebrandt G, Stienen MN. Sentinel Headache: A Warning Sign Preceding Every Fourth Aneurysmal Subarachnoid Hemorrhage. AJNR Am J Neuroradiol. 2015 Sep;36(9):E62-3. doi: 10.3174/ajnr.A4467. Epub 2015 Jul 16. No abstract available. PMID 26185328
- See also: Study synopsis — https://research.kssg.ch/Projekte/53442